CLINICAL TRIAL: NCT03697330
Title: Liberal Versus Restrictive Fluid Protocols in Adults Patients Undergoing Unilateral Orthopedic Lower Limb Surgery Under Spinal Anesthesia
Brief Title: Liberal Versus Restrictive Fluid Protocols in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, RAGAA AHMED HERDAN, lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Liberal Vs Restrictive Fluid
Record Dates: First submitted 2018-04-14; First posted 2018-10-05 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Intraoperative Complications
Keywords: liberal, restrictive, fluid, RIFLE
MeSH Terms: conditions — Intraoperative Complications | interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: comparing the effect of two different protocols of fluid therapy (liberal versus restrictive) in adult patients undergoing unilateral orthopedic lower limb surgery under spinal anesthesia
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done using computer generated table of random numbers in a 1:1 ratio and will be conducted using sequentially numbered, opaque and sealed envelope. The trial will be planned that neither the doctors (investigators) nor the patients will be aware of the group allocation and amount of fluid received. Intraoperative and postoperative data collections will be achieved by the same blinded anesthiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringer's lactate 18-20 ml/kg (Active Comparator): Patients will be randomly allocated into two groups of 40 patients each:
  Group L:will receive 18-20 ml/kg/h of Ringer's lactate starting from conduction of spinal anesthesia.
  Interventions: Drug: Ringer lactate
- Ringer's lactate 4-6 ml/kg (Active Comparator): Patients will be randomly allocated into two groups of 40 patients each:
  Group R: will receive 4-6 ml/kg/h of Ringer's lactate starting from conduction of spinal anesthesia.
  Interventions: Drug: Ringer lactate

INTERVENTIONS:
Drug: Ringer lactate — Randomization will be done using computer generated table of random numbers in a 1:1 ratio and will be conducted using sequentially numbered, opaque and sealed envelope. The trial will be planned that neither the doctors (investigators) nor the patients will be aware of the group allocation and amount of fluid received. Intraoperative and postoperative data collections will be achieved by the same blinded anesthiologist.
  Patients will be randomly allocated into two groups:
  Group L: 40 patients who will be subjected to ''liberal" approach of intraoperative 18-20 ml/kg/h of Ringer's lactate starting from conduction of spinal anesthesia.
  Group R: 40 patients who will be subjected to ''restrictive" approach of intraoperative 4-6 ml/kg/h of Ringer's lactate starting from conduction of spinal anesthesia.
  Blood loss will be replaced if more than 500 ml in a ratio of 3 ml crystalloid: 1 ml blood.
  Other Names: lactated ringers solution

SUMMARY:
The term acute kidney injury (AKI) is used to describe a rapid deterioration (hours to days) of renal function. This rapid deterioration leads to accumulation of plasma waste products, such as urea and creatinine.

Accumulation of urea and other nitrogen-containing substances in the blood stream lead to a number of symptoms, such as fatigue, loss of appetite, headache, nausea and vomiting. Marked increases in the potassium level can lead to irregularities in the heartbeat, which can be severe and life-threatening. Fluid balance is frequently affected, though blood pressure can be high, low or normal. Pain in the flanks may be encountered in some conditions (such as thrombosis of the renal blood vessels or inflammation of the kidney); this is the result of stretching of the fibrous tissue capsule surrounding the kidney.

Perioperative AKI is a leading cause of morbidity and mortality; It is associated with increased risk of sepsis, anemia, coagulopathy, and mechanical ventilation.

The first publication of consensus criteria for AKI was published in 2004. The system was named RIFLE (risk, injury, failure, loss of kidney function and end-stage renal failure) and used sCr or urine output to define AKI.

Later, in 2007, a modified definition of the RIFLE criteria was published by the Acute Kidney Injury Network (AKIN) .Although the AKIN criteria evolved from the RIFLE criteria, a major advance was the understanding that even small changes in sCr concentrations are associated with increased morbidity and mortality. The AKIN criteria allowed definition of AKI even without knowledge of baseline sCr.

In 2012, a clinical practice guideline of AKI was proposed by the Kidney Disease Improving Global Outcomes (KDIGO) Foundation. The guideline included a comprehensive review of AKI definition, risk assessment, diagnosis, prevention, treatment and renal replacement therapy.

A common practice to maintain effective blood volume and thus kidney perfusion is intravenous (I.V.) hydration. Correcting hypovolemia is an essential perioperative hemodynamic goal and appropriate hydration is considered important for the avoidance of AKI.

Perioperative fluid therapy has been studied extensively, but the optimal strategy remains controversial and uncertain. Much of the current debate surrounds the type of fluids administered (colloid versus crystalloid), the total volume administered (restrictive versus liberal), and whether the administration of fluids should be guided by hemodynamic goals (goal directed [GD] versus not goal directed).

Administering a large amount of I.V. fluid in the perioperative period is a common clinical practice. Although fluid loading may expand intravascular space, improve organ perfusion or tissue oxygenation and reduce minor postoperative complications in laparoscopic surgery, excessive fluid may also increase some perioperative complications.

Intraoperative urine output is often monitored but rarely responds to fluid administration. Clearance of fluid during general anesthesia is only a small fraction of that observed in conscious volunteers. Infusion of crystalloids during anesthesia shows reduced clearance and slower distribution such that intraoperative oliguria may not reflect fluid status or predict future AKI.

Given that liberal fluid administration can be correlated with worse postoperative outcome, the recommendation to maintain urine output of at least 0.5 ml/kg/h should be considered.

DETAILED DESCRIPTION:
Prior to surgery, all patients will undergo pre-anesthetic checkup including detailed history, physical, systemic examination, height and weight of the patient. All patients will be investigated for exclusion of any of the above mentioned contraindications. Routine preoperative laboratory investigations as complete blood count, grouping, coagulation profile, electrolytes and preoperative baseline serum creatinine will be measured. Patients should have low molecular weight heparin administered till the evening prior to daytime trauma lists. This precaution allows for an appropriate window of time to minimize the risk of bleeding related to neuraxial anesthesia. All patients will be kept nil per mouth 6 h for solids and 2 h for water and clear liquids.

Preparation of the patient and conduct of anesthesia:

Written consent and emergency resuscitation equipments including airway devices, advanced life support drugs for LA toxicity and intraoperative adverse events will be available. All patients will be anesthetized by the same team of anesthesiologists and operated upon by the same surgeon who will be unaware of the study medications.

After arriving at the operative room, the pulse oximetry, electrocardiography, temperature probe and non-invasive blood pressure monitor will be applied. A large bore I.V. cannula (18 gauge) will be inserted.

Spinal anesthesia will be used for all patients. Under aseptic technique and local skin infiltration with 1% lidocaine, spinal anesthesia will be performed at the L3-4 or L4-5 spinal interspace by 25 gauge spinal needle. After successful cerebrospinal fluid recognition, 10 mg heavy bupivacaine 0.5% mixed with 25 ug fentanyl will be injected into the subarachnoid space. Then the spinal needle will be removed and the patients will be positioned carefully to the suitable position. Once adequate anesthesia to at least T10 dermatome achieved, the operation will be allowed to be started. Supplemental oxygen will be administered via face mask at flow rate between 5 and 8 L/min. Management of the patients will be performed by another anesthesiologist unaware about the used protocol. Vital signs including heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressur (MBP) and arterial oxygen saturation (SpO2) will be recorded as baseline 5 min before conduction of spinal anesthesia, immediately after conduction of anesthesia then every 5 min till end of surgery. The level of sensory block will be assessed before beginning of surgery using an ice cube. Urinary catheter will be inserted for all patients. Hypotension defined as decrease in mean blood pressure (MAP) to more than 20% of baseline values will be treated with a 3 mg I.V. bolus of ephedrine repeated every 2 min if hypotension persists. If hypotension persists after 30 mg ephedrine, additional amounts of Ringer's lactate (5ml/ kg) will be infused through the 18 gauge cannula.

Patients will be asked to report any intraoperative pain or discomfort using visual analog scale (VAS) of 0-10.

After finishing surgery, patients will be transferred to the surgical ICU where they will be monitored by an intensivist who will be blinded to the study group.

Once the patients sent to ICU, both groups will receive 1.5 ml/kg/h of Ringer's lactate solution as fluid maintenance. Follow-up will be done for 5 days postoperatively using:

* Monitors for HR, SBP, DBP, MBP, SpO2 , respiratory rate and recovery time of motor blockade (up to Bromage 2)
* Analgesia: paracetamol 1 gm/ 6 hours regularly
* Supplemental oxygen will be provided in the first 24 hours after the operation if arterial oxygen saturation < 94%.
* Early mobilization: will improve oxygenation and respiratory function.
* Fluid balance as hypovolemia is common postoperatively and oral fluid intake should be encouraged over the intravenous route.
* Urinary tract infections (UTI): is common and urinary catheters should be removed as soon as possible to reduce the risk of infection and urine output will be collected and calculated as [after 12 hours, on day 2 (in 24 hours), 3 (in 24 hours), and 5 (in 24 hours after surgery]
* Routine laboratory investigations as CBC, coagulation profile, electrolytes, blood urea and serum creatinine.
* Symptoms suggestive of AKI: fatigue, loss of appetite, headache, nausea, vomiting and pain in the flanks Patients will be discharged from ICU when hemodynamics are stable and laboratory investigations are within normal.

ELIGIBILITY:
Inclusion Criteria:

Adults 18-50 years scheduled for unilateral orthopedic lower limb surgery

* ASA I and II
* Gender: both

Exclusion Criteria:

* Patient refusal
* Hypersensitivity to any local anesthetics
* Bleeding diathesis
* Skin lesions or wounds at the puncture site of the proposed block
* Psychiatric disorders
* Failed intra-thecal anesthesia or inadequate sensory block for surgery requiring conversion to general anesthesia
* Pregnancy
* Chronic kidney disease
* Diabetes mellitus, chronic heart, lung or liver disease
* Hemodynamic instability (intra and/or post-operative)
* Burn injury, usage of x-ray contrast and sepsis.
* Morbid obesity
* Corticosteroid usage

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
serum creatinine | 5 days postoperative
  mg/dl
urine output | 5 days postoperative
  ml

SECONDARY OUTCOMES:
SBP, DBP, MAP | 24 hours
  systolic blood pressure (mmHg) diastolic blood pressure (mmHg) mean arterial blood pressure (mmHg)
arterial oxygen saturation | 24 hours
heart rate | 24 hours
  beats/min

CONTACTS AND LOCATIONS:
Overall Officials: ragaa herdan, lecturer, Principal Investigator — Assiut University, Faculty of Medicine
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No